CLINICAL TRIAL: NCT06065670
Title: A Randomized, Double-Blind, Delayed Treatment, Placebo-Controlled Trial to Assess the Changes in Multi-parametric MRI in Patients With Acute Demyelinating Lesions Taking Clemastine Fumarate as a Myelin Repair Therapy
Brief Title: Assessing Changes in Multi-parametric MRI in Patients With Acute Demyelinating Lesions Taking Clemastine Fumarate as a Myelin Repair Therapy
Acronym: ReINFORCE
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-38525
Record Dates: First submitted 2023-09-19; First posted 2023-10-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Demyelinating Diseases; Demyelination; Corpus Callosum; Multiple Sclerosis Brain Lesion; Multiple Sclerosis Acute and Progressive; Clinically Isolated Syndrome, CNS Demyelinating
Keywords: acute brain lesions; mri; brain; demyelinating lesions; spinal cord
MeSH Terms: conditions — Demyelinating Diseases; Marchiafava-Bignami Disease | interventions — Clemastine; Sugars

STUDY DESIGN:
Intervention Model Description: This is a 6-month randomized double-blinded, placebo-controlled, delayed treatment study examining clemastine fumarate as a remyelinating agent in participants with multiple sclerosis. This trial will include n = 44 patients with a confirmed diagnosis of acute demyelinating lesions.
  Patients who fulfill the enrollment criteria will be randomly assigned (1:1) via block randomization using a random number generator to receive either clemastine for 90 days followed by placebo for 90 days (Clemastine 12 mg for 14 days, clemastine 8 mg for 76 days, then Placebo) or placebo for 90 days followed by clemastine for 90 days (Placebo, then Clemastine 12 mg for 14 days, the clemastine 8 mg for 76 days).
  If they are on one, patients will be permitted to remain on their standard disease-modifying treatment during the course of the study. These therapies have no identified effect on remyelination.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Clemastine 12 mg, then clemastine 8 mg, then Placebo (Experimental): Group 1 will receive the treatment (clemastine) for the first 90 days. They will receive clemastine 12 mg for 14 days followed by clemastine 8 mg for 76 days, and then switch to the placebo (a sugar pill) for the remaining 90 days
  Interventions: Drug: Clemastine Fumarate; Drug: Placebo
- Placebo, then Clemastine 12 mg, then Clemastine 8 mg (Experimental): Group 1 will receive the placebo for the first 90 days. Then, they will switch to clemastine (treatment) for 90 days. They will receive clemastine 12 mg for 14 days followed by clemastine 8 mg for the remaining 76 days.
  Interventions: Drug: Clemastine Fumarate; Drug: Placebo

INTERVENTIONS:
Drug: Clemastine Fumarate — 12 or 8 mg Clemastine tablet. Clemastine fumarate was approved by the Food and Drug Administration (FDA) for the treatment of allergic rhinitis (seasonal allergies) in 1977 and was approved for over-the-counter marketing in 1992. Clemastine is not FDA approved as a remyelinating therapy
  Other Names: Clemastine; Dayhist; Dayhist Allergy
Drug: Placebo — Matched sugar tablet
  Other Names: Sugar pill

SUMMARY:
The clinical trial is intended to assess for clinical evidence of Clemastine Fumarate as a myelin repair therapy in patients with acute inflammatory injury-causing demyelination as measured by multi-parametric MRI assessments.

No reparative therapies exist for the treatment of acute demyelinating lesions. Clemastine fumarate was identified along with a series of other antimuscarinic medications as a potential remyelinating agent using the micropillar screen (BIMA) developed at the University of California, San Francisco (UCSF). Following in vivo validation, an FDA IND exemption was granted to investigate clemastine for the treatment of multiple sclerosis in the context of chronic optic neuropathy. That pilot study was recently completed and is the first randomized control trial documenting efficacy for a putative remyelinating agent for the treatment of MS. The preselected primary efficacy endpoint (visual evoked potential) was met and a strong trend to benefit was seen for the principal secondary endpoint assessing function (low contrast visual acuity). That trial number was 13-11577.

This study seeks to follow up on that study and examine clemastine fumarate's protective and reparative effects in the context of acute demyelinating brain lesions as imaged by multi-parametric MRI assessments. The investigators will be assessing the effects of clemastine fumarate as a remyelinating therapy and assessing its effect on MRI metrics of lesions found in patients with a confirmed diagnosis of acute inflammatory injury-causing demyelination.

In addition to using conventional multi-parametric MRI assessments, this study will also evaluate a new MRI technique called Ultrashort Echo Time (UTE) MRI to assess the effects of clemastine fumarate as a remyelinating therapy of acute lesions found in patients with a confirmed diagnosis of acute inflammatory injury-causing demyelination and compare it to the other assessments.

DETAILED DESCRIPTION:
Treatments capable of remyelination are a major unmet need for demyelinating diseases that involve myelin damage, loss, or dysfunction in the central nervous system (CNS). Acute demyelination of axons is believed to be injurious to neurons and serves as a major contributor to irreversible cell loss that underlies permanent disability. Available treatments are primarily immunosuppressing, without directly addressing or fully preventing axonal degeneration and disability. Clemastine fumarate was identified along with a series of other antimuscarinic medications as a potential remyelinating agent using the micropillar screen (BIMA) developed at UCSF. The screen demonstrated that clemastine promoted the differentiation of the endogenous oligodendrocyte precursor cells (OPCs) into mature myelinating oligodendrocytes. Following in vivo validation, an FDA investigational new drug (IND) exemption was granted to investigate clemastine for the treatment of multiple sclerosis in the context of chronic optic neuropathy. That pilot study was recently completed and is the first randomized control trial documenting efficacy for a putative remyelinating agent for the treatment of MS. The preselected primary efficacy endpoint (visual evoked potential) was met and a strong trend to benefit was seen for the principal secondary endpoint assessing function (low contrast visual acuity). That trial number was 13-11577.

This clinical trial is intended to assess magnetic resonance imaging evidence of remyelination using Clemastine Fumarate in patients with acute demyelinated lesions. Specifically speaking, the primary objective will assess various multi-parametric MRI sequences on the corpus callosum region, a region that animal models studies identified as a promising candidate for assessing remyelination. The aim was to help define the potential for MRI in measuring remyelination in acute lesions, determine the optimal sequences and location for measuring myelin recovery, and help guide trial design for future remyelinating trials. Finally, the study is designed to assess tolerability and clinical efficacy of Clemastine using outcomes intended to assess for (a) adverse events and (b) recovery of myelin.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained prior to any assessment being performed.
* Patients diagnosed with relapsing remitting multiple sclerosis and a disease duration of < 15 years
* Male or female patients aged 18-55 years (inclusive)
* Use of appropriate contraception during period of trial (women). Before entry women must be:

  * Post-menopausal for at least 1 year OR
  * Surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, male partner vasectomy or otherwise incapable of pregnancy) OR
  * Practicing a highly effective method of birth control if sexually active, including hormonal prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double barrier method (e.g., condoms, diaphragm or cervical cap with spermicidal foam, cream or gel), or male partner sterilization consistent with local regulations regarding use of birth control methods for patients participating in clinical trials, for the duration of their participation in the study OR
  * Not heterosexually active (patients who are not heterosexually active at screening must agree to utilize a highly effective method of birth control if they become heterosexually active during their participation in the study) OR
  * Practicing true abstinence (when this is in line with the preferred and usual lifestyle of the subject) Period abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) is not an acceptable method.

Exclusion Criteria:

* Radiologic identification of marked brain atrophy relative to patients age based on recent MRI and interpretation of expert neuroradiologist or PI
* New lesion in most recent MRI (within 3 months)
* Hypersensitivity to clemastine or other arylalkylamine antihistamines, or any of the excipients.
* Treatment with corticosteroids within 30 days prior to screening.
* Expanded Disability Status Scale (EDSS) ≥ 4.5
* History of significant cardiac conduction block.
* History of cancer.
* Suicidal ideation or behavior in 6 months prior to baseline.
* Pregnancy, breastfeeding or planning to become pregnant.
* Involved with other study protocols simultaneously without prior approval.
* Concomitant use of any other putative remyelinating therapy as determined by the investigator.
* Prior treatment with total lymphoid irradiation, T cell or T cell receptor vaccination.
* Prior treatment with alemtuzumab, mitoxantrone, or cyclophosphamide.
* Serum creatinine > 1.5 mg/dL; aspartate transaminase (AST), alanine transaminase (ALT), or alkaline phosphatase > 2 times the upper limit of normal. (Reported within 72 hours)
* History of drug or alcohol abuse within the past year.
* Untreated B12 deficiency (as determined by B12 serological assessments and metabolites including methylmalonic acid [MMA] and homocysteine) or untreated hypothyroidism.
* Clinically significant cardiac, metabolic, hematologic, hepatic, immunologic, urologic, endocrinologic, neurologic, pulmonary, psychiatric, dermatologic, allergic, renal, or other major diseases that in the PI's judgment may affect the interpretation of study results or patient safety.
* History of or presence of clinically significant medical illness or laboratory abnormality that, in the opinion of the investigator would preclude participation in the study
* Inability to participate in MRI, including extreme claustrophobia.
* Any dental braces or permanent or undetachable metals in the jaw or face.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Corpus Callosum Myelin Water Fraction | This will be assessed at the baseline visit.
  The efficacy of clemastine relative to placebo at increasing the myelin water fraction (MWF) (measured in %) from magnetic resonance imaging of the corpus callosum.
Change from Baseline in Corpus Callosum Myelin Water Fraction at 3 Months | This will be assessed at the baseline and 3 month visits.
  The efficacy of clemastine relative to placebo at increasing the myelin water fraction (MWF) (measured in %) from magnetic resonance imaging of the corpus callosum. Change = (3-month % - Baseline %)
Change from Baseline in Corpus Callosum Myelin Water Fraction at 6 Months | This will be assessed at the baseline and 6 month visits.
  The efficacy of clemastine relative to placebo at increasing the myelin water fraction (MWF) (measured in %) from magnetic resonance imaging of the corpus callosum. Change = (6-month % - Baseline %)
Corpus Callosum T1 Relaxation Time | This will be assessed at the baseline visit.
  The efficacy of clemastine relative to placebo at shortening the T1 relaxation time (measured in seconds) within the corpus callosum using T1 mapping protocols in an MRI.
Change from Baseline in Corpus Callosum T1 Relaxation Time at 3 Months | This will be assessed at the baseline and 3-month visits.
  The efficacy of clemastine relative to placebo at shortening the T1 relaxation time (measured in seconds) within the corpus callosum using T1 mapping protocols in an MRI. (3-month time - Baseline time)
Change from Baseline in Corpus Callosum T1 Relaxation Time at 6 Months | This will be assessed at the baseline and 6-month visits.
  The efficacy of clemastine relative to placebo at shortening the T1 relaxation time (measured in seconds) within the corpus callosum using T1 mapping protocols in an MRI. (6-month time - Baseline time)
Corpus Callosum UTE Fraction | This will be assessed at the baseline visit.
  The efficacy of clemastine relative to placebo at increasing the ultrashort echo time (UTE) fraction (measured in %) derived from magnetic resonance imaging of the corpus callosum.
Change from Baseline in Corpus Callosum UTE Fraction at 3 Months | This will be assessed at the baseline and 3-month visits.
  The efficacy of clemastine relative to placebo at increasing the ultrashort echo time (UTE) fraction (measured in %) derived from magnetic resonance imaging of the corpus callosum. Change = (3-month % - Baseline %)
Change from Baseline in Corpus Callosum UTE Fraction at 6 Months | This will be assessed at the baseline and 6-month visits.
  The efficacy of clemastine relative to placebo at increasing the ultrashort echo time (UTE) fraction (measured in %) derived from magnetic resonance imaging of the corpus callosum. Change = (6-month % - Baseline %)

SECONDARY OUTCOMES:
Optic Radiation Myelin Water Fraction | This will be assessed at the baseline visit.
  The efficacy of Clemastine relative to placebo at increasing the MWF (measured in %) of the optic radiation.
Change from Baseline in Optic Radiation Myelin Water Fraction at 3 Months | This will be assessed at the baseline and 3-month visits.
  The efficacy of Clemastine relative to placebo at increasing the MWF (measured in %) of the optic radiation. Change = (3-month % - Baseline %)
Change from Baseline in Optic Radiation Myelin Water Fraction at 6 Months | This will be assessed at the baseline and 6-month visits.
  The efficacy of Clemastine relative to placebo at increasing the MWF (measured in %) of the optic radiation. Change = (6-month % - Baseline %)
Corticospinal Tract Myelin Water Fraction | This will be assessed at the baseline visit.
  The efficacy of clemastine relative to placebo at increasing the MWF (measured in %) of the corticospinal tract.
Change from Baseline in Corticospinal Tract Myelin Water Fraction at 3 Months | This will be assessed at the baseline and 3-month visits.
  The efficacy of clemastine relative to placebo at increasing the MWF (measured in %) of the corticospinal tract. (3-month % - Baseline %)
Change from Baseline in Corticospinal Tract Myelin Water Fraction at 6 Months | This will be assessed at the baseline and 6-month visits.
  The efficacy of clemastine relative to placebo at increasing the MWF (measured in %) of the corticospinal tract. (6-month % - Baseline %)
Optic Radiation T1 Relaxation time | This will be assessed at the baseline visit.
  To evaluate the efficacy of Clemastine relative to placebo at increasing the T1 relaxation time (measured in seconds) of the optic radiation.
Change from Baseline in Optic Radiation T1 Relaxation time at 3 Months | This will be assessed at the baseline and 3-month visits.
  To evaluate the efficacy of Clemastine relative to placebo at increasing the T1 relaxation time (measured in seconds) of the optic radiation. (3-month time - Baseline time)
Change from Baseline in Optic Radiation T1 Relaxation time at 6 Months | This will be assessed at the baseline and 6-month visits.
  To evaluate the efficacy of Clemastine relative to placebo at increasing the T1 relaxation time (measured in seconds) of the optic radiation. (6-month time - Baseline time)
Corticospinal Tract T1 Relaxation Time | This will be assessed at the baseline visit.
  To evaluate the efficacy of Clemastine relative to placebo at increasing the T1 relaxation time (measured in seconds) of the corticospinal tract.
Change from Baseline in Corticospinal Tract T1 Relaxation Time at 3 Months | This will be assessed at the baseline and 3-month visits.
  To evaluate the efficacy of Clemastine relative to placebo at increasing the T1 relaxation time (measured in seconds) of the corticospinal tract. (3-month time - Baseline time)
Change from Baseline in Corticospinal Tract T1 Relaxation Time at 6 Months | This will be assessed at the baseline and 6-month visits.
  To evaluate the efficacy of Clemastine relative to placebo at increasing the T1 relaxation time (measured in seconds) of the corticospinal tract. (6-month time - Baseline time)
Optic radiation UTE Fraction | This will be assessed at the baseline visit.
  The efficacy of clemastine relative to placebo at increasing the UTE fraction (measured in %) of the optic radiation.
Change from Baseline in Optic radiation UTE Fraction at 3 Months | This will be assessed at the baseline and 3-month visits.
  The efficacy of clemastine relative to placebo at increasing the UTE fraction (measured in %) of the optic radiation. Change = (3-month % - Baseline %)
Change from Baseline in Optic radiation UTE Fraction at 6 Months | This will be assessed at the baseline and 6-month visits.
  The efficacy of clemastine relative to placebo at increasing the UTE fraction (measured in %) of the optic radiation. Change = (6-month % - Baseline %)
Corticospinal Tract UTE Fraction | This will be assessed at the baseline visit.
  The efficacy of clemastine relative to placebo at increasing the UTE fraction (measured in %) of the corticospinal tract.
Change from Baseline in Corticospinal Tract UTE Fraction at 3 Months | This will be assessed at the baseline and 3-month visits.
  The efficacy of clemastine relative to placebo at increasing the UTE fraction (measured in %) of the corticospinal tract. (3-month % - Baseline %)
Change from Baseline in Corticospinal Tract UTE Fraction at 6 Months | This will be assessed at the baseline and 6-month visits.
  The efficacy of clemastine relative to placebo at increasing the UTE fraction (measured in %) of the corticospinal tract. (6-month % - Baseline %)
Lesion of interest (LOI) MWF | This will be assessed at the baseline visit.
  The efficacy of clemastine relative to placebo at increasing MWF (measured in %) of the lesion(s) of interest, stratified based on enhancement status on prior MRIs.
Change from Baseline in Lesion of interest (LOI) MWF at 3 Months | This will be assessed at the baseline and 3-month visits.
  The efficacy of clemastine relative to placebo at increasing MWF (measured in %) of the lesion(s) of interest, stratified based on enhancement status on prior MRIs. Change = (3-month % - Baseline %)
Change from Baseline in Lesion of interest (LOI) MWF at 6 Months | This will be assessed at the baseline and 6-month visits.
  The efficacy of clemastine relative to placebo at increasing MWF (measured in %) of the lesion(s) of interest, stratified based on enhancement status on prior MRIs. Change = (6-month % - Baseline %)
LOI T1 Relaxation Time | This will be assessed at the baseline visit.
  The efficacy of clemastine relative to placebo at increasing T1 relaxation time (measured in seconds) of the lesion(s) of interest, stratified based on enhancement status on prior MRIs.
Change from Baseline in LOI T1 Relaxation Time at 3 Months | This will be assessed at the baseline and 3-month visits.
  The efficacy of clemastine relative to placebo at increasing T1 relaxation time (measured in seconds) of the lesion(s) of interest, stratified based on enhancement status on prior MRIs. Change = (3-month time - Baseline time)
Change from Baseline in LOI T1 Relaxation Time at 6 Months | This will be assessed at the baseline and 6-month visits.
  The efficacy of clemastine relative to placebo at increasing T1 relaxation time (measured in seconds) of the lesion(s) of interest, stratified based on enhancement status on prior MRIs. Change = (6-month time - Baseline time)
LOI UTE Fraction | This will be assessed at the baseline visit.
  The efficacy of clemastine relative to placebo at increasing UTE fraction (measured in %) of the lesion(s) of interest, stratified based on enhancement status on prior MRIs.
Change from Baseline in LOI UTE Fraction at 3 Months | This will be assessed at the baseline and 3-month visits.
  The efficacy of clemastine relative to placebo at increasing UTE fraction (measured in %) of the lesion(s) of interest, stratified based on enhancement status on prior MRIs. Change = (3-month % - Baseline %)
Change from Baseline in LOI UTE Fraction at 6 Months | This will be assessed at the baseline and 6-month visits.
  The efficacy of clemastine relative to placebo at increasing UTE fraction (measured in %) of the lesion(s) of interest, stratified based on enhancement status on prior MRIs. Change = (6-month % - Baseline %)
Whole Brain MWF | This will be assessed at the baseline visit.
  The efficacy of clemastine relative to placebo at increasing MWF (measured in %) across the whole-brain divided into regions of normal-appearing white matter (NAWM), cortical gray matter, and deep gray matter.
Change from Baseline in Whole Brain MWF at 3 Months | This will be assessed at the baseline and 3-month visits.
  The efficacy of clemastine relative to placebo at increasing MWF (measured in %) across the whole-brain divided into regions of normal-appearing white matter (NAWM), cortical gray matter, and deep gray matter. Change = (3-month % - Baseline %)
Change from Baseline in Whole Brain MWF at 6 Months | This will be assessed at the baseline and 6-month visits.
  The efficacy of clemastine relative to placebo at increasing MWF (measured in %) across the whole-brain divided into regions of normal-appearing white matter (NAWM), cortical gray matter, and deep gray matter. Change = (6-month % - Baseline %)
Whole Brain T1 Relaxation Time | This will be assessed at the baseline visit.
  The efficacy of clemastine relative to placebo at increasing T1 relaxation time (measured in seconds) across the whole-brain divided into regions of normal-appearing white matter (NAWM), cortical gray matter, and deep gray matter.
Change from Baseline in Whole Brain T1 Relaxation Time at 3 Months | This will be assessed at the baseline and 3-month visits.
  The efficacy of clemastine relative to placebo at increasing T1 relaxation time (measured in seconds) across the whole-brain divided into regions of normal-appearing white matter (NAWM), cortical gray matter, and deep gray matter. (3-month time - Baseline time)
Change from Baseline in Whole Brain T1 Relaxation Time at 6 Months | This will be assessed at the baseline and 6-month visits.
  The efficacy of clemastine relative to placebo at increasing T1 relaxation time (measured in seconds) across the whole-brain divided into regions of normal-appearing white matter (NAWM), cortical gray matter, and deep gray matter. (6-month time - Baseline time)
Whole Brain UTE Fraction | This will be assessed at the baseline visit.
  The efficacy of clemastine relative to placebo at increasing the UTE fraction (measured in %) across the whole-brain divided into regions of normal-appearing white matter (NAWM), cortical gray matter, and deep gray matter.
Change from Baseline in Whole Brain UTE Fraction at 3 Months | This will be assessed at the baseline and 3-month visits.
  The efficacy of clemastine relative to placebo at increasing the UTE fraction (measured in %) across the whole-brain divided into regions of normal-appearing white matter (NAWM), cortical gray matter, and deep gray matter. Change = (3-month % - Baseline %)
Change from Baseline in Whole Brain UTE Fraction at 6 Months | This will be assessed at the baseline and 6-month visits.
  The efficacy of clemastine relative to placebo at increasing the UTE fraction (measured in %) across the whole-brain divided into regions of normal-appearing white matter (NAWM), cortical gray matter, and deep gray matter. Change = (6-month % - Baseline %)
Clemastine Tolerability | This will be assessed at the baseline visit.
  The tolerability of Clemastine in this population. This will include a special focus with regards to fatigue as this is a major symptom for patients suffering from demyelinating lesions using the Fatigue Scale for Motor and Cognitive Functions (FSMC). The FSMC is scored from 1 through 5 for each question. A high score of 100 indicates a high level of fatigue. The lowest score, 20, indicates low level of fatigue.
Change from Baseline in Clemastine Tolerability at 3 Months | This will be assessed at the baseline and 3-month visits.
  The tolerability of Clemastine in this population. This will include a special focus with regards to fatigue as this is a major symptom for patients suffering from demyelinating lesions using the Fatigue Scale for Motor and Cognitive Functions (FSMC). The FSMC is scored from 1 through 5 for each question. A high score of 100 indicates a high level of fatigue. The lowest score, 20, indicates low level of fatigue. Change = (3-month tolerability - Baseline tolerability)
Change from Baseline in Clemastine Tolerability at 6 Months | This will be assessed at the baseline and 6-month visits.
  The tolerability of Clemastine in this population. This will include a special focus with regards to fatigue as this is a major symptom for patients suffering from demyelinating lesions using the Fatigue Scale for Motor and Cognitive Functions (FSMC). The FSMC is scored from 1 through 5 for each question. A high score of 100 indicates a high level of fatigue. The lowest score, 20, indicates low level of fatigue. Change = (6-month tolerability - Baseline tolerability)

CONTACTS AND LOCATIONS:
Overall Officials: Ari J Green, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Sandler Neurosciences Building, Neurological Clinical Research Unit, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mei F, Fancy SPJ, Shen YA, Niu J, Zhao C, Presley B, Miao E, Lee S, Mayoral SR, Redmond SA, Etxeberria A, Xiao L, Franklin RJM, Green A, Hauser SL, Chan JR. Micropillar arrays as a high-throughput screening platform for therapeutics in multiple sclerosis. Nat Med. 2014 Aug;20(8):954-960. doi: 10.1038/nm.3618. Epub 2014 Jul 6. PMID 24997607
- [Background] Marques JP, Kober T, Krueger G, van der Zwaag W, Van de Moortele PF, Gruetter R. MP2RAGE, a self bias-field corrected sequence for improved segmentation and T1-mapping at high field. Neuroimage. 2010 Jan 15;49(2):1271-81. doi: 10.1016/j.neuroimage.2009.10.002. Epub 2009 Oct 9. PMID 19819338
- [Background] Sheth V, Shao H, Chen J, Vandenberg S, Corey-Bloom J, Bydder GM, Du J. Magnetic resonance imaging of myelin using ultrashort Echo time (UTE) pulse sequences: Phantom, specimen, volunteer and multiple sclerosis patient studies. Neuroimage. 2016 Aug 1;136:37-44. doi: 10.1016/j.neuroimage.2016.05.012. Epub 2016 May 5. PMID 27155128
- [Background] Green AJ, Gelfand JM, Cree BA, Bevan C, Boscardin WJ, Mei F, Inman J, Arnow S, Devereux M, Abounasr A, Nobuta H, Zhu A, Friessen M, Gerona R, von Budingen HC, Henry RG, Hauser SL, Chan JR. Clemastine fumarate as a remyelinating therapy for multiple sclerosis (ReBUILD): a randomised, controlled, double-blind, crossover trial. Lancet. 2017 Dec 2;390(10111):2481-2489. doi: 10.1016/S0140-6736(17)32346-2. Epub 2017 Oct 10. PMID 29029896
- [Background] Gagliardo A, Galli F, Grippo A, Amantini A, Martinelli C, Amato MP, Borsini W. Motor evoked potentials in multiple sclerosis patients without walking limitation: amplitude vs. conduction time abnormalities. J Neurol. 2007 Feb;254(2):220-7. doi: 10.1007/s00415-006-0334-5. Epub 2007 Feb 17. PMID 17308868